CLINICAL TRIAL: NCT00002542
Title: Double-Blind Randomized Trial of Tamoxifen Versus Placebo in Patients With Node Positive or High Risk Node Negative Breast Cancer Who Have Completed CMF, CEF, or AC Adjuvant Chemotherapy
Brief Title: Tamoxifen in Treating Women With High-Risk Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA12; CAN-NCIC-MA12; NCI-V93-0323; CDR0000063224 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Doxorubicin; Epirubicin; Fluorouracil; Methotrexate; Tamoxifen; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Drug: tamoxifen citrate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen. Chemotherapy uses different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase III trial to study the effectiveness of tamoxifen following surgery and chemotherapy in treating women who have stage I breast cancer at high risk of recurrence or stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the duration of overall survival and disease-free survival in premenopausal women with operable, high risk node negative or axillary node-positive breast cancer who have undergone complete surgical resection of all known disease by means of total or partial mastectomy, and have received standard adjuvant chemotherapy with cyclophosphamide, methotrexate, and fluorouracil (CMF), cyclophosphamide, epirubicin, and fluorouracil (CEF), or doxorubicin and cyclophosphamide (AC) followed by either daily tamoxifen for 5 years or placebo. II. Compare the short- and long-term toxicity in patients receiving tamoxifen versus placebo. III. Monitor follicle-stimulating hormone, luteinizing hormone, and estradiol levels, and determine whether overall survival and disease-free survival are affected by hormonal or menopausal status during or at completion of adjuvant chemotherapy or during or after tamoxifen or placebo treatment in these patients.

OUTLINE: This is a randomized, double blind study. Patients are stratified by adjuvant chemotherapy regimen (cyclophosphamide, epirubicin, and fluorouracil vs cyclophosphamide, methotrexate, and fluorouracil vs cyclophosphamide and doxorubicin), hormone receptor status (ER and/or PR positive vs ER and PR negative), number of positive nodes (1-3 vs 4-9 vs 10 or more), and participating institution. Patients receive one of three regimens of adjuvant chemotherapy at the discretion of the investigator. Regimen A: Patients receive oral cyclophosphamide on days 1-14 and epirubicin IV and fluorouracil IV on days 1 and 8. Courses repeat every 28 days for a total of 6 courses. Following chemotherapy, lumpectomy patients receive local radiotherapy daily for 5 weeks. Regimen B: Patients receive oral cyclophosphamide on days 1-14 or cyclophosphamide IV on day 1 and 8, methotrexate on days 1 and 8, and fluorouracil IV on days 1 and 8. Courses repeat every 28 days for a total of 6 courses. Concurrent with or following chemotherapy, lumpectomy patients receive local radiotherapy daily for 5 weeks. Regimen C: Patients receive doxorubicin IV and cyclophosphamide IV every 21 days for a total of 4 courses. Following chemotherapy, lumpectomy patients receive local radiotherapy daily for 5 weeks. Patients are then randomized to receive either oral tamoxifen or a placebo once daily for 5 years, beginning within 6 weeks of completion of chemotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Adenocarcinoma of the breast with 1 or more histologically proven positive axillary nodes OR Adenocarcinoma of the breast with negative axillary nodes or adverse prognostic factors such that the patient is at high risk for recurrence and node negative lesion is characterized by the following features: Tumor at least 1 cm Poorly differentiated, SBR grade III, or MSBR grade V and/or lymphatic/vascular invasion Pathologic review by experienced breast pathologist recommended if grade is unspecified and lymphatic/vascular invasion is absent Disease considered potentially curable and treated by 1 of the following: Complete surgical removal of the breast plus axillary node dissection Partial surgical removal of the breast plus axillary node dissection, with the intention of giving breast irradiation following completion of an adjuvant chemotherapy regimen Regional nodal or chest wall irradiation not prohibited but strongly discouraged No evidence of residual tumor in the axilla following dissection No microscopic evidence of residual tumor at the resection margins following total mastectomy Further excision highly recommended if there is microscopic residual disease present at partial mastectomy margins If further excision is not undertaken, a radiotherapy boost to the tumor bed is required in addition to breast irradiation given following protocol chemotherapy Disease clinically staged prior to surgery as T1-T3a, N0-2, M0 No clinical T4 disease, i.e.: No extension to the chest wall No edema (including peau d'orange) No skin ulceration No satellite skin nodules confined to the same breast No inflammatory carcinoma Disease pathologically staged following surgery as TNM stage I, II, or III (T0-4; N0-2; M0) T4 allowed only with dermal involvement on pathology assessment No evidence of metastatic disease beyond the homolateral axillary nodes on pre-chemotherapy chest x-ray, bone scan (with radiographs of suspicious areas), and abdominal ultrasound (required only if bilirubin, alkaline phosphatase, or AST/ALT are elevated) Simultaneous bilateral breast carcinoma allowed Complete tumor resection on both breasts required Axillary dissection on both sides must meet criteria as above if both sides are clinically node-positive Axillary dissection on the second side optional if the axilla is clinically negative at the time of surgery and the other side is node-positive Adjuvant chemotherapy must begin within 14 weeks of initial pathologic diagnosis Hormone receptor status: Any receptor level allowed (values must be available if biochemical method used; immunocytochemical assay permitted)

PATIENT CHARACTERISTICS: Age: Not specified Sex: Female Menopausal status: Pre- or perimenopausal, i.e., meeting at least 1 of the following criteria: Normal menstruation Amenorrhea for less than 1 year (up to 3 years in patients under age 52) Biochemical evidence of ovarian function Hysterectomy without bilateral oophorectomy in patients under age 56 Premenopausal women no greater than age 50 who were started on replacement hormone therapy before amenorrhea are eligible Performance status: ECOG 0-2 prior to chemotherapy Hematopoietic: WBC at least 3,000/mm3 Polymorphs and bands at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: (unless abdominal ultrasound indicates liver metastasis) Alkaline phosphatase no greater than 2 times normal AST and/or ALT no greater than 2 times normal Renal: Not specified Other: No history of serious underlying medical illness or psychiatric or addictive disorder No second malignancy within 5 years except: Curatively treated nonmelanomatous skin cancer Curatively treated endometrium, colon, or thyroid cancer or carcinoma in situ of the cervix No plan for pregnancy during the 5-year study period Fertile women must use effective contraception (other than oral contraception) Accessible for treatment and follow-up

PRIOR CONCURRENT THERAPY: Biologic therapy: Colony-stimulating factors allowed (use must be documented) Chemotherapy: No prior chemotherapy No concurrent other cytotoxic therapy Endocrine therapy: Adjuvant tamoxifen (20 mg po daily) allowed up to 2 weeks before or during adjuvant chemotherapy provided drug is discontinued at randomization No long-term prednisone or other hormones Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 1993-07-20 (Actual); Primary Completion 2007-03-07 (Actual); Study Completion 2011-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivien HC Bramwell, MB, BS, PhD, FRCP, Study Chair — London Health Sciences Centre
Locations (48):
- Canada (48):
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - The Royal Victoria Hospital, Barrie
  - William Osler Health Centre, Brampton Memorial, Brampton
  - Tom Baker Cancer Centre, Calgary
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown
  - Cross Cancer Institute, Edmonton
  - Regional Cancer Program of the Hopital Regional, Greater Sudbury
  - QEII Health Sciences Center, Halifax
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton
  - Centre Hospitalier Regional de Lanaudiere, Joliette
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston
  - L'Hotel-Dieu de Levis, Lévis
  - London Regional Cancer Program, London
  - Credit Valley Hospital, Mississauga
  - CHUM - Hopital Notre-Dame, Montreal
  - McGill University - Dept. Oncology, Montreal
  - CHUM - Hotel Dieu du Montreal, Montreal
  - CHUM - Pavillon Saint-Luc, Montreal
  - Stronach Regional Health Centre at Southlake, Newmarket
  - Lakeridge Health Oshawa, Oshawa
  - Ottawa Health Research Institute - General Division, Ottawa
  - Penticton Regional Hospital, Penticton
  - Peterborough Regional Health Centre, Peterborough
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec
  - CHA-Hopital Du St-Sacrement, Québec
  - University Institute of Cardiology and, Québec
  - Allan Blair Cancer Centre, Regina
  - Atlantic Health Sciences Corporation, Saint John
  - Saskatoon Cancer Centre, Saskatoon
  - Algoma District Cancer Program, Sault Ste. Marie
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke
  - Niagara Health System, St. Catharines
  - BCCA - Fraser Valley Cancer Centre, Surrey
  - Thunder Bay Regional Health Science Centre, Thunder Bay
  - Toronto East General Hospital, Toronto
  - Odette Cancer Centre, Toronto
  - St. Michael's Hospital, Toronto
  - Mount Sinai Hospital, Toronto
  - Univ. Health Network-The Toronto General Hospital, Toronto
  - Univ. Health Network-Princess Margaret Hospital, Toronto
  - Women's College Hospital, Toronto
  - St. Joseph's Health Centre, Toronto
  - Trillium Health Centre - West Toronto, Toronto
  - Humber River Regional Hospital, Toronto
  - BCCA - Vancouver Cancer Centre, Vancouver
  - BCCA - Vancouver Island Cancer Centre, Victoria
  - Windsor Regional Cancer Centre, Windsor
  - CancerCare Manitoba, Winnipeg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bramwell VHC, Pritchard KI, Tu D, et al.: How compliant are patients with oral hormonal therapies? Data from a randomized, placebo controlled study of tamoxifen after adjuvant chemotherapy in premenopausal women with early breast cancer (NCIC CTG MA.12). [Abstract] Breast Cancer Res Treat 106 (1): A-3055, 2007.
- [Result] Bramwell VH, Pritchard KI, Tu D, et al.: Tamoxifen (T) compared to placebo (P), after adjuvant chemotherapy (CT), in premenopausal women with early breast cancer (EBC): interim results of NCIC-CTG MA.12. [Abstract] J Clin Oncol 25 (Suppl 18): A-547, 2007.